CLINICAL TRIAL: NCT06331546
Title: Gastrointestinal Oxalate Absorption in Calcium Oxalate Stone Disease
Brief Title: Gut Oxalate Absorption in Calcium Oxalate Stone Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sonia Fargue, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB300004693-GIA; R01DK137784 (NIH)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Kidney Stone; Kidney Calculi; Urolithiasis; Urolithiasis, Calcium Oxalate; Nephrolithiasis; Nephrolithiasis, Calcium Oxalate; Oxalate Urolithiasis; Oxaluria; Healthy
MeSH Terms: conditions — Kidney Calculi; Urolithiasis; Nephrolithiasis, Calcium Oxalate; Nephrolithiasis; Hyperoxaluria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Idiopathic Calcium Oxalate Kidney Stone Patients (Experimental): Low and High oxalate fixed diets. Soluble oxalate absorption test.
  Interventions: Dietary Supplement: Low-oxalate diet; Dietary Supplement: High-oxalate diet; Other: soluble oxalate gut absorption test
- Healthy non-kidney stone forming individuals (Active Comparator): Low and High oxalate fixed diets. Soluble oxalate absorption test.
  Interventions: Dietary Supplement: Low-oxalate diet; Dietary Supplement: High-oxalate diet; Other: soluble oxalate gut absorption test

INTERVENTIONS:
Dietary Supplement: Low-oxalate diet — 4 days of fixed eucaloric diet with low oxalate (<60 mg/day), normal calcium content (600-1000 mg/day)
Dietary Supplement: High-oxalate diet — 4 days of fixed eucaloric diet with moderately high oxalate (250-300 mg/day), normal calcium content (600-1000 mg/day)
Other: soluble oxalate gut absorption test — Oral ingestion of 13C2-oxalate and sucralose.

SUMMARY:
The goal of this clinical trial study is to test if patients with idiopathic calcium oxalate kidney stones have an increased absorption of dietary oxalate, which would lead to increased urinary excretion of oxalate.

The study will recruit adult patients with a history of calcium oxalate kidney stones and healthy volunteers without kidney stones.

Participants will

* ingest fixed diets containing low and moderately high amounts of oxalate for 5 days at a time
* ingest a soluble form of oxalate and sugar preparations to test gut permeability
* collect urine, blood, stool and breath sample during the fixed diets and the soluble oxalate test

DETAILED DESCRIPTION:
In this study the investigators propose to measure the net gastrointestinal absorption of oxalate both by food-bound oxalate, using low- (<60 mg/day) and high- (250-300 mg/day) oxalate diets (600-800 mg daily calcium in both), and by the soluble 13C2-oxalate oral test in both Calcium Oxalate Kidney Stone patients and matched controls.

Phase 1. Screening and low-oxalate diet 24-hr urinary excretions. Between the University of Alabama at Birmingham (UAB) and the University of Texas Southwestern Medical Center (UTSW), the study will enroll 40 subjects with idiopathic Calcium Oxalate Kidney Stone (20 Males/20 Females) and 40 non-kidney stone forming controls (20 Males/20 Females). Participants in the two groups will be matched for age (within 10 yrs) and gender. Screening will include blood complete metabolic profile and two 24-hr urine specimens collected at home on self-choice diets and anthropometric measurements.

Participants will then ingest the controlled low-oxalate (<60 mg/d) diet for 5 consecutive days and collect two 24-hr urines after 2 days of dietary equilibration.

Phase 2. 13C2-Oxalate gut absorption tests. On Day 5, participants will arrive after an overnight fast in the research unit to undergo the 13C2-oxalate absorption test. After a 1-hour baseline urine collection, they will ingest an oral load containing 100 mg 13C2-oxalate and 1 g sucralose, dissolved in bottled water. For the next 9 hrs, blood and urine will be collected hourly, and breath as more time points. They will remain on the fixed diet for 24 hrs with a breakfast 2 hours after the load, lunch 6 hrs post-load, and dinner at home 12 hrs post-load. They will collect the remainder of their 24-hr urine at home and the totality of the stool eliminated during the first 24 hrs after the load using kits provided.

Phase 3. High-oxalate diet 24-hr urinary excretions. After a minimum of 1 week wash-out period, during which participants will eat freely, participants will consume the high oxalate (250-300 mg/day) diet for the next 4 days. Two 24-hr urine specimens will be collected after 2 days of equilibration and a fasting blood draw on the morning of Day 5.

.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 yrs
* Body Mass Index > 18.5 kg/m2
* Normal fasting serum electrolytes on comprehensive metabolic profile
* Willing to ingest fixed diets
* Willing to stop supplements (vitamins including vitamin C, calcium (citrate or carbonate) and other minerals, herbal supplements, nutritional aids, probiotics) for 2 weeks before start and during study.
* For stone formers: first time or recurrent Calcium Oxalate stone former. Composition of most recent stone ≥ 50% calcium oxalate if available, uric acid component <20%

Exclusion Criteria:

* Chronic Kidney Disease stage 4-5
* Primary hyperoxaluria, Enteric (secondary) hyperoxaluria
* Liver, bowel, endocrine or renal diseases (other than idiopathic Calcium Oxalate kidney stones) or any other condition that may influence the absorption, transport or urinary excretion of ions, which will compromise the interpretation of results, including: Cystic fibrosis, Celiac disease, Cystinuria, Uric acid stone former, Nephrotic syndrome, Sarcoidosis, Renal tubular acidosis, Primary hyperparathyroidism, Neurogenic bladder, Urinary diversion, Chronic diarrhea, Bariatric surgery, Inflammatory bowel disease
* Pregnancy or breast-feeding
* Incompatible dietary requirements with the study, food allergies or intolerance to any of the foods in study menus
* Active malignancy or treatment for malignancy within 12 months prior to screening
* Utilization of immunosuppressive medication
* Uncontrolled hypertension or diabetes
* Diabetes type 1
* Chronic NSAID use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — all
Enrollment: 80 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Net Gastrointestinal absorption of food-bound oxalate | 4 day
  difference between 24-hour urinary oxalate excretion on the high oxalate diet and the low oxalate diet, normalized to the difference in dietary oxalate composition of the two diets (%)

SECONDARY OUTCOMES:
Absorption of soluble 13C2-oxalate | 1 day
  Proportion of 13C2-oxalate recovered in urine to the amount orally ingested (%)
Estimated endogenous oxalate synthesis (oxalate mg/day) | 2 days
  24-hour urinary oxalate excretion on the low oxalate diet (mg/day)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Fargue, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UTSW, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No